CLINICAL TRIAL: NCT00688402
Title: A Double-blind, Randomized, Cross-over Design, Phase 1 Pharmacodynamic Study to Investigate the Effect of Different Formulations of AZD3355 for the Development of Paresthesiae After Dosing in Healthy Subjects
Brief Title: Study to Compare Different Formulations of AZD3355
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Debra G. Silberg, MD, PhD, Medical Science Director, AZD3355, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D9120C00031; EudraCT nr 2007-007126-22
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Reflux Inhibitor; GERD; formulations
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — lesogaberan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): IR Formulation 65 mg
  Interventions: Drug: AZD3355
- 2 (Experimental): IR Formulation 150 mg
  Interventions: Drug: AZD3355
- 3 (Experimental): MR formulation, 1h 65 mg
  Interventions: Drug: AZD3355
- 4 (Experimental): MR Formulation, 1h 150 mg
  Interventions: Drug: AZD3355
- 5 (Experimental): MR Formulation, 2h 150 mg
  Interventions: Drug: AZD3355

INTERVENTIONS:
Drug: AZD3355 — Single dose
  Other Names: Lesogaberan

SUMMARY:
The purpose of the study is to compare different formulations of AZD3355 in regard to possible adverse events such as sensations of numbness, tinglings and heat in the skin.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Female subjects with no childbearing potentials or using highly efficient contraceptive methods
* Clinically normal physical findings

Exclusion Criteria:

* Clinically significant illness within 2 weeks prior to the first dose of investigational product
* History of clinically significant disease
* Use of prescribed medication during the 2 weeks before administration of the first dose of investigational product

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Specific AE questions | During 0-4 hours post dose

SECONDARY OUTCOMES:
PK variables | Frequent sampling up to 36 hours post dose
Safety variables (other adverse events, blood pressure, pulse, safety lab) | During the whole treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ersdal, PhD, Study Director — AstraZeneca R&D, Mölndal, Sweden; Aslak Rautio, MD, Principal Investigator — Quintiles Hermelinen, Varvsgatan 53, SE-972 33 Luleå, Sweden
Locations (1):
- Research Site, Varvsgatan, Lulea, Sweden